CLINICAL TRIAL: NCT00369044
Title: Chronic Administration of Prednisone in Management of Patients With Decompensated Congestive Heart Failure
Brief Title: Prednisone for Decompensated Congestive Heart Failure
Status: Suspended | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hebei Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 200608A
Record Dates: First submitted 2006-08-28; First posted 2006-08-29 (Estimated); Last update posted 2009-04-08 (Estimated); Status verified 2007-06

CONDITIONS: Heart Failure, Congestive
Keywords: decompensated heart failure; prednisone; diuretics; diuresis
MeSH Terms: conditions — Heart Failure | interventions — Prednisone

INTERVENTIONS:
Drug: prednisone

SUMMARY:
We designed this, randomized, double-blind, placebo-controlled trial to determine the clinical efficacy of chronic administration of prednisone on renal function and clinical status when added to standard care.

DETAILED DESCRIPTION:
Studies showed that glucocorticoids could specifically dilate renal vessel, increase in GFR, and regulate synthesis and release of atrial natriuretic peptide (ANP), upregulate ANP receptors on vascular endothelial cells, leading to significant diuresis and natriuresis. Adding glucocorticoids to standard care may potentiate the diuretic and natriuretic effects of diuretics and improve renal function, thus improve the clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized with primary diagnosis of CHF
* Patients with normal cortical function
* LVEF <40%
* Significant fluid overload, defined as ≥ 2 of the following

  * Enlarged liver or ascites
  * Peripheral or sacral edema ( ≥ 2+)
  * Jugular venous distention ≥ 10 cm
  * Pulmonary rales, pleural effusion on chest x-ray or orthopnea

Exclusion Criteria:

* Severe stenotic valvular disease
* Serum creatinine > 4 mg/dl
* Patient refusal
* Any signs of infection or any condition that would contraindicate an glucocorticoids use
* Poor controlled hypertension
* Poor controlled diabetes mellitus
* Active myocarditis
* Malignancy or other terminal illness

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-10; Study Completion 2008-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in serum creatinine level, Patient and physician-assessed symptom scales at day 1, day 3, the end of week 1 and week 2

SECONDARY OUTCOMES:
Daily urine volume, changes in body weight, serum electrolyte levels at the end of week 1, week 2, respectively, and overall safety profile

CONTACTS AND LOCATIONS:
Overall Officials: Kunshen Liu, MD, Principal Investigator — The First Hospital of Hebei Medical University
Locations (1):
- The First Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

REFERENCES:
- [Background] Liu C, Chen H, Zhou C, Ji Z, Liu G, Gao Y, Tian L, Yao L, Zheng Y, Zhao Q, Liu K. Potent potentiating diuretic effects of prednisone in congestive heart failure. J Cardiovasc Pharmacol. 2006 Oct;48(4):173-6. doi: 10.1097/01.fjc.0000245242.57088.5b. PMID 17086096